CLINICAL TRIAL: NCT02613182
Title: Open-label Extension Study to Evaluate the Long-term Safety and Tolerability of NEOD001 in Subjects With Light Chain (AL) Amyloidosis
Brief Title: Open-label Extension Study of NEOD001 in Subjects With Light Chain (AL) Amyloidosis
Acronym: OLE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: NEOD001 program terminated due to lack of clinical benefit
Sponsor: Prothena Biosciences Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEOD001-OLE001
Record Dates: First submitted 2015-11-18; First posted 2015-11-24 (Estimated); Results first posted 2019-05-16 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: AL Amyloidosis
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis | interventions — birtamimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open Label (Experimental): Open Label Study Drug NEOD001
  Interventions: Drug: NEOD001

INTERVENTIONS:
Drug: NEOD001 — NEOD001

SUMMARY:
The rationale for this study is to provide additional treatment with NEOD001 for subjects who complete Study NEOD001-001, and to continue to evaluate long term safety and tolerability. All subjects in the current NEOD001 trials are being dosed at 24 mg/kg, which will be continued in this study.

DETAILED DESCRIPTION:
The rationale for this study is to provide additional treatment with NEOD001 for subjects who complete Study NEOD001-001, and to continue to evaluate long term safety and tolerability. All subjects in the current NEOD001 trials are being dosed at 24 mg/kg, which will be continued in this study. The primary objective of the study is to evaluate long-term safety and tolerability of NEOD001 and the secondary objectives are to assess the immunogenicity of NEOD001 and to incorporate serum NEOD001 concentrations in a population pharmacokinetic (PK) analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Previously enrolled and treated for at least 9 months in Study NEOD001-001
2. Ability to understand and willingness to sign an informed consent form prior to initiation of any study procedures
3. Has adequate bone marrow reserve, hepatic and renal function, as demonstrated by:

   * Absolute neutrophil count (ANC) ≥1.0 ×109/L
   * Platelet count ≥75 × 109/L
   * Hemoglobin ≥9 g/dL
   * Total bilirubin ≤2 times the upper limit of normal (× ULN)
   * Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) ≤3 × ULN
   * Estimated glomerular filtration rate ≥30 mL/minute
4. Seated systolic blood pressure 90 to 180 mmHg
5. ECOG Performance Status 0 to 2
6. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 28 days prior to the first administration of study drug and agree to use highly effective physician-approved contraception from 30 days prior to the first study drug administration to 90 days following the last study drug administration
7. Male subjects must be surgically sterile or must agree to use highly effective physician-approved contraception from 30 days prior to the first study drug administration to 90 days following the last study drug administration

Exclusion Criteria:

1. Any new medical contraindication or clinically significant abnormality on physical, neurological, laboratory, vital signs, or electrocardiogram (ECG) examination (e.g., atrial fibrillation; with the exception of subjects for whom the ventricular rate is controlled) that precludes continued or initiation of treatment with NEOD001 or participation in the study
2. History of Grade ≥3 infusion-associated adverse events (AEs) or hypersensitivities to NEOD001 or any of its excipients
3. Treatment with any anticancer therapy (standard or investigational) within the 14 days prior to the first dose of study drug. In addition, subjects must have fully recovered (i.e., National Cancer Institute Common Terminology Criteria for Adverse Events [CTCAE] Grade 1 [exception: subjects with prior bortezomib may have CTCAE Grade 2 neuropathy]) from the clinically significant toxic effects of that treatment
4. Received any of the following within the specified time frame prior to the first administration of study drug:

   * Hematopoietic growth factors, transfusions of blood or blood products within 1 week
   * Major surgery within 2 weeks
   * Radiotherapy within 2 weeks
   * Transplant within 8 weeks
   * Investigational drug other than NEOD001 within 4 weeks
   * Another experimental anti-amyloid therapy other than NEOD001 within 2 years
5. Uncontrolled symptomatic orthostatic hypotension
6. Myocardial infarction, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia, within 6 months prior to the first dose of study drug
7. Uncontrolled infection
8. Secondary malignancy, with the exception of:

   * Adequately treated basal cell carcinoma, squamous cell carcinoma, or in situ cervical cancer
   * Adequately treated stage I cancer from which the subject is currently in remission
   * Any other cancer from which the subject has been disease-free for ≥3 years
9. Uncontrolled human immunodeficiency virus (HIV), hepatitis B, or hepatitis C infection
10. Women who are lactating

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-02; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Stanford Cancer Institute (SCI), Stanford, California
  - Tufts Medical Center, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- NEOD001 24 mg/kg: NEOD001, 24 mg/kg IV every 28 days for 22 months
Period: Overall Study
Arm/Group | NEOD001 24 mg/kg
Started | 34
Number of Patients Dosed | 34
Completed | 0
Not Completed | 34
Not completed — Death | 6
Not completed — Physician Decision | 1
Not completed — Study Terminated by Sponsor | 21
Not completed — Withdrawal by Subject | 6

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- NEOD001 24 mg/kg: NEOD001, 24 mg/kg IV every 28 days for 22 months (open-label study drug)
Arm/Group | NEOD001 24 mg/kg
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.1 (8.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 34
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 1
  White | 32
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Long-term Safety and Tolerability of NEOD001
Description: Adverse events are defined as any unfavorable and unintended diagnosis, symptom, sign (including an abnormal laboratory finding), syndrome, or disease which either occurs during study, having been absent at baseline, or, if present at baseline, appears to worsen. Serious adverse events are any untoward medical occurrences that result in death, are life threatening, require (or prolong) hospitalization, cause persistent or significant disability/incapacity, result in congenital anomalies or birth defects, or are other conditions which in judgment of investigators represent significant hazards.
Time Frame: From initiation of study drug through the last study visit or up to 30 days after date of last dose, whichever came first, assessed up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | NEOD001 24 mg/kg
Number analyzed (Participants) | 34
Participants
  Overall number of baseline subjects | 34
  Serious Adverse Events | 12
  Non-Serious Adverse Events | 34
  Death (all causes) | 6
  Death (from Adverse Events) | 1

ADVERSE EVENTS:
Time Frame: Initiation of study drug through the last study visit or up to 30 days after date of last dose
Description: AE that newly appears, increases in frequency, or worsens in severity following initiation of study
Groups:
- NEOD001 24 mg/kg: 24 mg/kg IV every 28 days for 22 months
Arm/Group | NEOD001 24 mg/kg
All-Cause Mortality (participants affected / at risk) | 6/34
Serious Adverse Events (participants affected / at risk) | 12/34
Other Adverse Events (participants affected / at risk) | 34/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NEOD001 24 mg/kg (N=34)
Infection (Infections and infestations) | 1 — Respiratory syncytial virus infection
Lung Infection (Infections and infestations) | 1
Respiratory syncytial virus infection (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Cardiac failure (Cardiac disorders) | 2
Acute myocardial infarction (Cardiac disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1
Hypervolaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Asthenia (General disorders) | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Hypotension (Vascular disorders) | 1
Viral pharyngitis (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NEOD001 24 mg/kg (N=34)
Upper respiratory tract infection (Infections and infestations) | 15
Urinary tract infection (Infections and infestations) | 3
Pneumonia (Infections and infestations) | 2
Oedema peripheral (Gastrointestinal disorders) | 9
Fatigue (General disorders) | 6
Pyrexia (General disorders) | 3
Chest discomfort (General disorders) | 2
Constipation (Gastrointestinal disorders) | 8
Diarrhoea (Gastrointestinal disorders) | 6
Abdominal pain (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 5
Abdominal distension (Gastrointestinal disorders) | 3
Abdominal discomfort (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 2
Eructation (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Weight increased (Investigations) | 3
Blood creatine phosphokinase increased (Investigations) | 2
Blood creatinine increased (Investigations) | 2
Weight decreased (Investigations) | 2
Contusion (Injury, poisoning and procedural complications) | 4
Fall (Injury, poisoning and procedural complications) | 3
Infusion related reaction (Injury, poisoning and procedural complications) | 2
Dizziness (Nervous system disorders) | 5
Headache (Nervous system disorders) | 3
Ecchymosis (Skin and subcutaneous tissue disorders) | 6
Rash (Skin and subcutaneous tissue disorders) | 3
Anaemia (Blood and lymphatic system disorders) | 4
Neutropenia (Blood and lymphatic system disorders) | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 3
Decreased appetite (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Insomnia (Psychiatric disorders) | 7
Hypertension (Vascular disorders) | 3
Hypotension (Vascular disorders) | 2
Palpitations (Cardiac disorders) | 2
Dysuria (Renal and urinary disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI, institution and the sponsor have agreed that the PI and institution may publish or disclose study results from their site after the earlier of (a) publication of the complete multicenter study results or (b) 18 months after database lock for the multicenter study. The sponsor has at least 45 days to review a proposed publication and may request deletion of confidential information and up to 60 days additional delay to obtain patent protection.

DOCUMENTS (2):
  • Study Protocol (2017-03-09): https://cdn.clinicaltrials.gov/large-docs/82/NCT02613182/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-14): https://cdn.clinicaltrials.gov/large-docs/82/NCT02613182/SAP_001.pdf